CLINICAL TRIAL: NCT00921388
Title: Exercise for Smoking Cessation in Postmenopausal Women
Brief Title: Exercise or Relaxation for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-097-2; 1R01DA024872-01A1 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Nicotine Dependence; Smoking Cessation
Keywords: Smoking Cessation; Exercise; Postmenopausal women; CHANTIX; varenicline
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Motor Activity | interventions — Varenicline; Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise program
  Interventions: Other: Varenicline and smoking cessation counseling; Behavioral: Exercise or relaxation treatment
- 2 (Other): Relaxation program
  Interventions: Other: Varenicline and smoking cessation counseling

INTERVENTIONS:
Other: Varenicline and smoking cessation counseling — All subjects receive smoking cessation counseling and varenicline 0.5mg daily for three days then twice a day for the next four days; then 1 mg twice a day for 11 weeks. Counseling is integrated within the exercise or relaxation treatment program.
  Other Names: CHANTIX
Behavioral: Exercise or relaxation treatment — One hour exercise sessions twice a week for 8 weeks, then once a week for 8 weeks, then once every other week for 4 weeks. Subjects in the control group receive a relaxation program that controls for contact time.
  Other Names: exercise program
  Arms: 1

SUMMARY:
This research study is being done to find out if adding a moderate exercise program or a relaxation program to a smoking cessation treatment program will improve smoking cessation and health in postmenopausal women. We hope to learn which group is more successful at quitting, has less symptoms of withdrawal from smoking and has improved health.

DETAILED DESCRIPTION:
Prevalence of smoking among women has declined more slowly in women than among men. Women who quit smoking substantially reduce the risk of premature death. A multi-modal approach to smoking cessation with combined behavioral and pharmacological interventions generally yields the highest success rates. The majority of subjects who are able to achieve abstinence return to smoking. Smoking relapse rates are 50-80% within one year with the majority of smokers relapsing within the first 3 months. Interventions are needed to both enhance smoking cessation rates and prevent relapse rates in order to substantially impact long-term quit rates.We intend to compare the effectiveness of a smoking cessation program combined with a moderate exercise program to an identical smoking cessation program combined with a relaxation-meditation control condition.

In a substudy, we will also evaluate the effectiveness of the intervention in premenopausal women (N=40)

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women at least 45 years of age
* Smoking at least 10 cigarettes per day
* Motivated to quit smoking
* Ambulatory
* Currently exercising for 90 minutes of moderate exercise or less per week
* Motivated to exercise
* Permission from Primary Care Provider
* Good general health

Exclusion Criteria:

* Denied medical clearance from primary care provider
* Unstable angina or uncompensated heart failure
* Systolic blood pressure greater than 165 or diastolic blood pressure greater than 100
* Heart attack or stroke within the preceding 6 months
* Hip fracture within the preceding 6 months
* Unstable medical or psychiatric disorder (e.g., current major depressive disorder or substance abuse or dependence)
* Exercise-exacerbated neuromuscular disorder
* Treatment for depression within the last year
* Estimated creatinine clearance of less than 30cc/minute
* Current use of a smoking cessation aid (i.e., bupropion, NRT, clonidine)
* Current use of psychotropic medication for a psychiatric problem
* Prescription narcotic abuse or dependence with the exception of people that have been stabilized on Methadone Maintenance or Suboxone
* Previous serious adverse event with Chantix use

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2009-03; Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
To evaluate whether adding an established moderate resistance/aerobic exercise program for postmenopausal women 45 years of age and older to a standard smoking cessation treatment program improves short and long term smoking outcomes. | Week 12 and Week 64

SECONDARY OUTCOMES:
To examine the main and interactive effects of history of depression and exercise on smoking cessation treatment. | Week 12 and Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Oncken, MD MPH, Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902